CLINICAL TRIAL: NCT02051114
Title: Discovering the Antecedents of Rheumatoid Arthritis Flare
Status: Active, not recruiting | Type: Observational
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Other Study IDs: DOR-0833
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Longitudinal study of patients with rheumatoid arthritis comparing measures of disease activity with blood samples.

DETAILED DESCRIPTION:
80% of patients living with rheumatoid arthritis can expect fluctuations in their symptoms over time. Dramatic increases in disease activity are considered flare. This study will follow patients with increased risk for flare prospectively for one year. Serial questionnaires and disease activity scores will be compared to blood samples to better understand the molecular phenotype of rheumatoid arthritis flares.

ELIGIBILITY:
Inclusion Criteria:

* 2010 criteria for Rheumatoid Arthritis
* Swelling of at least one joint and or elevated acute phase reactants
* Greater than or equal to 40 years old or less than or equal to 65 year old female sex
* cyclic citrullinated peptide antibody + in the past 12 months

Exclusion Criteria:

* hemoglobin < 9
* white blood cell count < 3.5
* Diagnosis of any active malignancy within the last 3 years besides non-melanomatous skin cancer
* Diagnosis of diabetes and requires insulin
* HIV+, Hep B S Ag+, Hep C polymerase chain reaction +
* Untreated latent tuberculosis
* Diagnosis of any additional systemic autoimmune connective tissue disease
* Inability to reliably complete study requirements
* History, physical, social or laboratory findings suggestive of any other medical or psychological condition that would, in the opinion of the principal investigator, make the candidate ineligible for the study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2014-02; Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
RNA transcripts that correlate with rheumatoid arthritis disease activity | 1 year
  Blood drawn at various times throughout one year will be correlated with fluctuations in RA disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Dana E Orange, MD, MS, Principal Investigator — The Rockefeller University Hospital
Locations (1):
- The Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Background] Orange DE, Yao V, Sawicka K, Fak J, Frank MO, Parveen S, Blachere NE, Hale C, Zhang F, Raychaudhuri S, Troyanskaya OG, Darnell RB. RNA Identification of PRIME Cells Predicting Rheumatoid Arthritis Flares. N Engl J Med. 2020 Jul 16;383(3):218-228. doi: 10.1056/NEJMoa2004114. PMID 32668112
- [Background] Brewer RC, Lanz TV, Hale CR, Sepich-Poore GD, Martino C, Swafford AD, Carroll TS, Kongpachith S, Blum LK, Elliott SE, Blachere NE, Parveen S, Fak J, Yao V, Troyanskaya O, Frank MO, Bloom MS, Jahanbani S, Gomez AM, Iyer R, Ramadoss NS, Sharpe O, Chandrasekaran S, Kelmenson LB, Wang Q, Wong H, Torres HL, Wiesen M, Graves DT, Deane KD, Holers VM, Knight R, Darnell RB, Robinson WH, Orange DE. Oral mucosal breaks trigger anti-citrullinated bacterial and human protein antibody responses in rheumatoid arthritis. Sci Transl Med. 2023 Feb 22;15(684):eabq8476. doi: 10.1126/scitranslmed.abq8476. Epub 2023 Feb 22. PMID 36812347